CLINICAL TRIAL: NCT07261800
Title: Sex-specific Differences in the Association Between Leg Fat and Diabetes Risk: The Mediating Role of Visceral Adipose Tissue
Brief Title: Sex-specific Differences in the Association Between Leg Fat and Diabetes Risk
Status: Completed | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xuan Song, Associated physician, Qianfoshan Hospital
Other Study IDs: S877
Record Dates: First submitted 2025-09-09; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus; Visceral Adipose Tissue; Body Fat Distribution
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetes group: Participants diagnosed with type 2 diabetes based on clinical guidelines, including elevated fasting plasma glucose (FPG) and/or HbA1c levels. This group will help assess how regional fat distribution (particularly leg-fat percentage) correlates with T2D risk.
  Interventions: Other: Not Applicable - Retrospective study
- non-diabetes group: Participants without T2DM, with normal glucose metabolism and no history of insulin resistance. This group is used as a reference for comparing the metabolic effects of adipose distribution with the T2DM group.
  Interventions: Other: Not Applicable - Retrospective study

INTERVENTIONS:
Other: Not Applicable - Retrospective study — Not Applicable - Retrospective study

SUMMARY:
This study investigates the association between LFP, VAT and T2DM using DXA in 542 adults. We apply penalized regression, generalized additive models (GAM), and causal mediation analysis to explore whether higher LFP reduces diabetes risk and whether this effect is mediated by VAT. Sex-specific analyses further clarify the biological differences in adipose distribution. The findings aim to improve understanding of fat distribution and metabolic health.

DETAILED DESCRIPTION:
T2DM is a major public health concern, and growing evidence suggests that not all body fat confers equal metabolic risk. Beyond total adiposity, the regional distribution of fat strongly influences insulin resistance and diabetes development. VAT is metabolically detrimental, promoting inflammation and lipotoxicity, whereas lower-body subcutaneous fat, particularly in the legs and gluteofemoral region, may exert protective metabolic effects by serving as a "safe storage" depot for excess lipids. However, the causal mechanisms underlying these associations remain incompletely understood, and whether the protective role of LFP differs by sex remains unclear.

This study aims to elucidate the metabolic and causal pathways linking LFP, VAT, and diabetes risk in adults. Using DXA for precise body composition assessment, the study evaluates the associations between LFP, VAT, and T2DM prevalence, with a focus on sex-specific effects. A total of 542 adult participants will be analyzed, including both men and women with and without T2DM. Clinical, biochemical, and anthropometric data will be collected concurrently.

The analytic framework integrates multiple complementary approaches:

1. Penalized regression models (LASSO, ridge, elastic net) will identify the most predictive adiposity components for T2DM while minimizing collinearity.
2. GAMs will examine potential nonlinear relationships between LFP, VAT, and diabetes risk, separately for male and female.
3. Causal mediation analysis will quantify the extent to which VAT mediates the relationship between LFP and diabetes, providing mechanistic insight into adipose redistribution pathways.
4. Inverse-probability-of-treatment weighting (IPTW) will strengthen causal inference by balancing covariates across LFP strata.
5. Two-sample Mendelian randomization (MR) will further test the causal effect of genetically predicted LFP on T2DM risk using summary-level genome-wide association data.

We hypothesize that higher LFP will be associated with lower diabetes risk and that this protective effect will be partially mediated by reduced VAT accumulation, particularly in females.

This study integrates imaging-based body composition, causal modeling, and genetic validation to bridge observational and causal evidence. The findings are expected to improve the understanding of sex-specific fat distribution in metabolic health and support the development of personalized prevention strategies targeting regional adiposity rather than total body fat.

ELIGIBILITY:
Inclusion Criteria:

Adults (≥18 years old)

Available DXA measurement of fat distribution

Complete fasting glucose or diabetes diagnosis record

Exclusion Criteria:

* Missing key variables (fat distribution, diabetes status)

Severe systemic disease interfering with data integrity

Implausible or inconsistent records

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who underwent DXA examination and had complete clinical and biochemical data.
Sampling Method: Non-Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of diabetes in relation to lower extremity fat | Baseline
  T2DM will be defined according to standard diagnostic criteria (fasting plasma glucose ≥ 7.0 mmol/L and/or HbA1c ≥ 6.5%, or a physician diagnosis). The primary outcome is the association between LFP and diabetes status, estimated using multivariable logistic regression and causal mediation analysis.

SECONDARY OUTCOMES:
Mediating Effect of VAT | baseline
  Quantification of the indirect effect of VAT in the association between LFP and T2DM risk, estimated via causal mediation analysis.
Sex-specific Differences in the LFP-T2D Association | Baseline
  Evaluation of whether the association between LFP and diabetes risk differs between males and females using sex-stratified models and interaction testing.

OTHER OUTCOMES:
Nonlinear Relationship Between LFP/VAT and T2D Risk (GAM Analysis) | baseline
  Characterization of potential nonlinear (threshold or saturation) relationships between LFP, VAT, and diabetes risk using generalized additive models (GAMs).
Causal Association Between Genetically Predicted LFP and T2D (Mendelian Randomization) | baseline
  Two-sample Mendelian randomization (MR) using genome-wide association study (GWAS) summary statistics to test the causal effect of genetically predicted LFP on T2D risk.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Song, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, China

IPD SHARING:
Plan to Share IPD: No